CLINICAL TRIAL: NCT05428137
Title: Randomized, Double Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of a Live and Heat Treated Bacteria Strain on Body Composition in Overweight Individuals
Brief Title: Study of Safety and Efficacy of a Probiotic and Postbiotic in Overweight Individuals
Acronym: KOBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCTB202014
Record Dates: First submitted 2022-05-24; First posted 2022-06-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Abdominal Obesity
MeSH Terms: conditions — Obesity; Obesity, Abdominal | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: 3 arm parallel design
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic (Active Comparator): Live bacteria strain in a form of a capsule daily for 16 weeks
  Interventions: Dietary Supplement: Probiotic
- Postbiotic (Active Comparator): Heat treated bacteria strain in a form of a capsule daily for 16 weeks
  Interventions: Dietary Supplement: Postbiotic
- Placebo (Placebo Comparator): Placebo in a form of a capsule administered for 16 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Live bacteria strain in a form of a capsule daily for 16 weeks
  Arms: Probiotic
Dietary Supplement: Postbiotic — Heat treated bacteria strain in a form of a capsule daily for 16 weeks
  Arms: Postbiotic
Other: Placebo — Placebo in a form of a capsule given for 16 weeks
  Arms: Placebo

SUMMARY:
Investigate the effect of a probiotic (live bacteria) and postbiotic (heat-treated bacteria) strains in overweight individuals.

DETAILED DESCRIPTION:
This study aims to investigate the safety and efficacy of live and heat treated bacteria on body composition of overweight individuals. The trial will be run in a single research centre and will recruit adult men and women, with BMI of 25-33kg/m2 with abdominal obesity.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25-33kg/m2
* Abdominal obesity (female waist circumference>85cm; male waist circumference>90cm)
* written informed consent

Exclusion Criteria:

* Taking the following medication within 1 month before starting the study: appetite stimulants/suppressants, lipid lowering drug, contraceptive
* taking antibiotics within 2 months before starting the study
* secondary obesity or secondary hypertension, diabetes type 1, GI disease, dyslipidaemia, type 2diabetes, hypertension
* consumption of pre- and probiotic-enriched products or dietary supplement for at least 4 weeks prior to the first screening visit
* nicotine, drug or alcohol abuse,
* other condition that, in the opinion of the investigators, would make participation not in the best interest of the patient or could prevent, limit or confound the Study's results

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in visceral fat area | From week 0 to Week 16
  Difference in visceral fat area (cm^2) measured using CT from week 0 to week 16

SECONDARY OUTCOMES:
Change in body weight | Week 0, Week 12, Week 16
  Body weight (kg) will be assessed at week 0, Week 12, Week 16
Change in waist circumference | Week 0, Week 12, Week 16
  Change in waist circumference (cm) at week 0, week 12 and week 16
Change in body fat composition | Week 0, Week 12, Week 16
  Change in body fat composition using dual-energy x-ray absorptiometry (DEXA) at week 0, Week 12, Week 16
Change in peripheral blood cholesterol | Week 0, Week 16
  Change in Cholesterol concentration (mg/dL) (total, HDL, LDL) in peripheral blood from week 0 to week 16
Change in serum insulin concentration | Week 0, Week 16
  Change in serum insulin from week 0 to week 16
Change in peripheral blood glucose | Week 0, Week 16
  Change in blood glucose from week 0 to week 16
Change in plasma leptin levels | Week 0, Week 16
  Change in leptin week 0 to week 16
Dietary survey | Week 0, Week 16
  Food cravings will be assessed using the Food Craving Questionnaires (FCQ) at week 0 and week 16. The change in score compared to baseline and between groups will be assessed at the end of the study.
Microbiome analysis | Week 0, Week 16
  Stool samples will be collected from participants to analyse change in intestinal microbiota community composition by 16SRNA sequencing
Mood questionnaire | Week 0, Week 16
  Participants mood will be assessed using the PHQ-9 (Patient Health Questionnaire-9). The change in score compared to baseline and between groups will be assessed at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ramon Vidal, Study Chair — ADM Biopolis
Locations (1):
- The Catholic University of Korea St. Vincent's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No